CLINICAL TRIAL: NCT00076219
Title: CSP #530 - Intensive vs. Conventional Renal Support in Acute Renal Failure
Brief Title: Acute Renal Failure Trial Network (ATN) Study
Acronym: ATN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 530
Record Dates: First submitted 2004-01-15; First posted 2004-01-19 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Acute Renal Failure
Keywords: Acute Renal Failure; Renal Replacement Therapy; multi-site randomization trial; Hemodialysis; Hemofiltration; Critical Illness; Hemodiafiltration
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive renal replacement therapy (Experimental): In the intensive management strategy, intermittent hemodialysis and sustained low-efficiency dialysis were provided 6 times per week, and continuous venovenous hemodiafiltration was provided at 35 mL/kg/hour.
  Interventions: Procedure: renal replacement therapy
- Less-intensive renal replacement therapy (Active Comparator): In the less-intensive management strategy, intermittent hemodialysis and sustained low-efficiency dialysis were provided 3 times per week, and continuous venovenous hemodiafiltration was provided at 20 mL/kg/hour.
  Interventions: Procedure: renal replacement therapy

INTERVENTIONS:
Procedure: renal replacement therapy — renal replacement therapy

SUMMARY:
This is a multi-center, prospective, randomized, parallel-group trial of an intensive strategy vs conventional strategy of renal replacement therapy for the treatment of acute renal failure secondary to acute tubular necrosis in critically ill patients. The primary hypothesis is that the intensive strategy will reduce 60-day all cause mortality by 10% compared to the conventional strategy - i.e.,a reduction from 55% in the conventional arm to 45% in the intensive arm. Secondary outcomes are 60-day in-hospital all-cause mortality, 1-year all cause mortality, and recovery of renal function by day 28. The study will recruit 1164 patients over a period of 3 years, 8 months and each patient will be actively followed for 60 days.

DETAILED DESCRIPTION:
Primary Hypothesis: An intensive management strategy for renal support in critically ill patients with acute renal failure decreases mortality as compared to less intensive (conventionally recommended) management strategies for renal replacement therapy.

Secondary Hypotheses: An intensive management strategy for renal support in critically ill patients with acute renal failure will shorten the duration of ARF, decrease the incidence and duration of non-renal complications and is cost-effective as compared to less intensive (conventionally recommended) management strategies for renal replacement therapy.

Primary Outcomes: 60-day all-cause mortality.

Secondary Outcomes: All-cause hospital mortality; 1-year all cause mortality; recovery of renal function; duration of renal support (dialysis-free days); ICU and hospital length of stay (ICU-and hospital-free days); non-renal organ system failures (organ-failure-free days); and discharge to "home" not on dialysis.

Study Abstract: The optimal management of renal replacement therapy (RRT) in acute renal failure (ARF) is uncertain. The VA/NIH Acute Renal Failure Trial Network (ATN Study) is designed to test the hypothesis that a strategy of intensive renal support will decrease mortality in critically ill patients with ARF as compared to less intensive (conventionally recommended) management. In this multicenter, prospective trial, patients with ARF due to acute tubular necrosis will be randomized equally to intensive or conventional management strategies for RRT.

In both arms, RRT will be initiated using the same criteria. Hemodynamically stable patients (SOFA cardiovascular score: 0-2) will receive intermittent hemodialysis (IHD) while hemodynamically unstable patients (SOFA cardiovascular score: 3-4) will be treated with continuous venovenous hemodiafiltration (CVVHDF) or sustained low-efficiency hemodialysis (SLED). Patients will convert between modalities of therapy as hemodynamic status changes over time. The intensity of therapy in IHD and SLED will vary between groups based on treatment frequency; with treatments provided 6-times per week in the intensive management strategy arm and 3-times per week in the conventional management strategy arm. In CVVHDF, intensity of therapy will vary based on effluent flow rate with a prescribed flow rate of 35 mL/kg/hour in the intensive management strategy arm and 20 mL/kg/hour in the conventional management strategy arm.

Protocol therapy will be continued until renal function recovers or until day 28. The primary study end-point will be 60-day all-cause mortality. Other end-points will include hospital and 1-year mortality, recovery of renal function, duration of renal support, ICU and hospital length of stay, hospital discharge off of dialysis and development/recovery of non-renal organ failure. An economic analysis will be performed to assess the costs and relative cost effectiveness of the two strategies.

The planned total enrollment of 1164 patients at 27 institutions over 44 months was selected to provide a power of 0.90 to detect a reduction in mortality from 55% to 45% with alpha=0.05 assuming a dropout/loss-to-follow-up rate of 10%.

Study enrollment began in November 2003 and closed after 44 months on July 2, 2007. Total enrollment was 1124 subjects. Fewer than 3% of subjects withdrew from protocol therapy. Follow-up for the primary study endpoint (60-day all-cause mortality) concluded on August 31, 2007; one-year follow-up will conclude in July 2008.

A type of dialysis solution used in the study was under IND with No. 67,631 and granted by Center for Drug Evaluation and Research in FDA.

ELIGIBILITY:
Inclusion Criteria:

* Acute renal failure clinically consistent with a diagnosis of acute tubular necrosis
* Plan for renal replacement therapy by clinical team
* Receiving care in a critical care unit
* One non-renal organ failure or sepsis
* Age 18 or older
* Patient or surrogate provides informed consent

Exclusion Criteria:

* Baseline serum creatinine > 2 mg/dL (177 mol/L) in males, > 1.5 mg/dL (133 mol/L) in females
* Acute renal failure clinically believed to be due to an etiology other than acute tubular necrosis
* More than 72 hours since meeting both of the following conditions:

  1. Fulfillment of the definition of ARF; and
  2. BUN > 100 mg/dL (36 mmol/L)
* More than 1 hemodialysis treatment or more than 24 hours since starting continuous renal replacement therapy
* Prior kidney transplant
* Pregnancy
* Prisoner
* Weight > 128.5 kg
* Non-candidacy for renal replacement therapy
* Moribund state
* Patient not expected to survive 28 days because of underlying terminal chronic medical condition
* Comfort-measures-only status
* Participation in a concurrent interventional study
* Patient/surrogate refusal
* Physician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1124 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Palevsky, Study Chair — VA Pittsburgh Health Care System
Locations (22):
- United States (22):
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Miami, Miami, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Result] Palevsky PM, O'Connor TZ, Chertow GM, Crowley ST, Zhang JH, Kellum JA; US Department of Veterans Affairs/National Institutes of Health Acute Renal Failure Trial Network. Intensity of renal replacement therapy in acute kidney injury: perspective from within the Acute Renal Failure Trial Network Study. Crit Care. 2009;13(4):310. doi: 10.1186/cc7901. Epub 2009 Aug 11. PMID 19678919
- [Result] Palevsky PM, O'Connor T, Zhang JH, Star RA, Smith MW. Design of the VA/NIH Acute Renal Failure Trial Network (ATN) Study: intensive versus conventional renal support in acute renal failure. Clin Trials. 2005;2(5):423-35. doi: 10.1191/1740774505cn116oa. PMID 16317811
- [Result] Johansen KL, Smith MW, Unruh ML, Siroka AM, O'Connor TZ, Palevsky PM; VA/NIH Acute Renal Failure Trial Network. Predictors of health utility among 60-day survivors of acute kidney injury in the Veterans Affairs/National Institutes of Health Acute Renal Failure Trial Network Study. Clin J Am Soc Nephrol. 2010 Aug;5(8):1366-72. doi: 10.2215/CJN.02570310. Epub 2010 May 27. PMID 20507953
- [Result] Joyce VR, Smith MW, Johansen KL, Unruh ML, Siroka AM, O'Connor TZ, Palevsky PM; Veteran Affairs/National Institutes of Health Acute Renal Failure Trial Network. Health-related quality of life as a predictor of mortality among survivors of AKI. Clin J Am Soc Nephrol. 2012 Jul;7(7):1063-70. doi: 10.2215/CJN.00450112. Epub 2012 May 17. PMID 22595826
- [Derived] Zampieri FG, Serpa-Neto A, Wald R, Bellomo R, Bagshaw SM; STARRT-AKI and RENAL Investigators. Hierarchical endpoints in critical care: A post-hoc exploratory analysis of the standard versus accelerated initiation of renal-replacement therapy in acute kidney injury and the intensity of continuous renal-replacement therapy in critically ill patients trials. J Crit Care. 2024 Aug;82:154767. doi: 10.1016/j.jcrc.2024.154767. Epub 2024 Mar 11. PMID 38461657
- [Derived] Kwong YD, Liu KD, Hsu CY, Cooper B, Palevsky PM, Kellum JA, Johansen KL, Miaskowski C. Subgroups of Patients with Distinct Health Utility Profiles after AKI. Kidney360. 2023 Jul 1;4(7):881-889. doi: 10.34067/KID.0000000000000201. Epub 2023 Jun 26. PMID 37357351
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Naorungroj T, Neto AS, Wang A, Gallagher M, Bellomo R. Renal outcomes according to renal replacement therapy modality and treatment protocol in the ATN and RENAL trials. Crit Care. 2022 Sep 6;26(1):269. doi: 10.1186/s13054-022-04151-5. PMID 36068554
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Sharma S, Kelly YP, Palevsky PM, Waikar SS. Intensity of Renal Replacement Therapy and Duration of Mechanical Ventilation: Secondary Analysis of the Acute Renal Failure Trial Network Study. Chest. 2020 Oct;158(4):1473-1481. doi: 10.1016/j.chest.2020.05.542. Epub 2020 May 26. PMID 32470389
- [Derived] Ng YH, Ganta K, Davis H, Pankratz VS, Unruh M. Vascular Access Site for Renal Replacement Therapy in Acute Kidney Injury: A Post hoc Analysis of the ATN Study. Front Med (Lausanne). 2017 Apr 11;4:40. doi: 10.3389/fmed.2017.00040. eCollection 2017. PMID 28443283

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Renal Replacement Therapy | Less-intensive Renal Replacement Therapy
Started | 563 | 561
Completed | 545 | 550
Not Completed | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Renal Replacement Therapy | Less-intensive Renal Replacement Therapy | Total
Number analyzed (Participants) | 563 | 561 | 1124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 341 | 335 | 676
  >=65 years | 222 | 226 | 448
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (15.3) | 59.7 (15.2) | 59.7 (15.3)
Gender [Number; unit: participants] — One subject has missing gender.
  participants
    Female | 154 | 176 | 330
    Male | 409 | 384 | 793

OUTCOME MEASURES:

1. Primary Outcome: 60-day All-cause Mortality
Description: 60-day all-cause mortality
Time Frame: 60 days
Population: Number of all-cause mortality by day 60
Measure: Number; unit: participants
Arm/Group | Intensive Renal Replacement Therapy | Less-intensive Renal Replacement Therapy
Number analyzed (Participants) | 563 | 561
participants | 302 | 289
Statistical Analysis 1: Comparison: Intensive Renal Replacement Therapy vs Less-intensive Renal Replacement Therapy; Test type: Superiority or Other; p = 0.47, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.86 to 1.40], Standard Error of Mean 0.12

ADVERSE EVENTS:
Arm/Group | Intensive Renal Replacement Therapy | Less-intensive Renal Replacement Therapy
Serious Adverse Events (participants affected / at risk) | 287/563 | 280/561
Other Adverse Events (participants affected / at risk) | 0/563 | 0/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Renal Replacement Therapy (N=563) | Less-intensive Renal Replacement Therapy (N=561)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 9 (9)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Electromechanical dissociation (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 9 (9)
Pericardial rub (Cardiac disorders) | 0 (0) | 1 (1)
Rhythm idioventricular (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 6 (8)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 3 (3)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 7 (7) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 3 (3) | 4 (4)
Chest pain (General disorders) | 0 (0) | 2 (3)
Death (General disorders) | 6 (6) | 2 (2)
Multi-organ failure (General disorders) | 40 (40) | 46 (48)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 9 (9) | 5 (5)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 1 (1)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Lung transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (3) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 3 (3) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 2 (2) | 2 (2)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 32 (34) | 33 (35)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 22 (22) | 31 (33)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of bone marrow transplant (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Non-accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anoxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 3 (3)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardiac operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Thoracotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Ventricular septal defect repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Air embolism (Vascular disorders) | 1 (2) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 2 (2)
Aortic dissection (Vascular disorders) | 0 (0) | 3 (3)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypoperfusion (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 58 (82) | 50 (78)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No